CLINICAL TRIAL: NCT01453335
Title: Utilizing a Near Infrared Vein Visualization Device To Increase Peripheral Intravenous Access Targets in Pediatric & Adult Patients (% Venous Options)
Brief Title: Percentage Venous Options in Pediatrics & Adults
Status: Completed | Type: Observational
Sponsor: Christie Medical Holdings, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP1001
Record Dates: First submitted 2011-08-23; First posted 2011-10-17 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Veins
Keywords: Veins; Catheter Segments; Vascular Access; VeinViewer Vision

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
VeinViewer® Vision will significantly increase the number of peripheral intravenous catheter access targets perceived by clinicians with experience in intravenous cannulation when compared to the number of access targets that these clinicians are able to visualize unaided or to palpate.

ELIGIBILITY:
Pediatric arm

Inclusion Criteria:

* Age 17 years of age or younger,
* Intact skin, without rash,irritation, scarring, open abrasion or other injury in these sites.
* Parent or guardian is English speaking
* Pediatric patients 8 years older will be asked to provide assent
* Participant does not have an acute or critical medical illness or injury requiring immediate evaluation and/or treatment.

Exclusion Criteria:

* 18 years of age or older
* No intact upper extremities
* Patient has had current or recent (within 6 months) venous access in the arm that will be evaluated.
* Acute or critical illness or injury requiring immediate or urgent evaluation and treatment.

Adult arm:

Inclusion Criteria:

* Age 18 years or older,
* At least one intact upper extremity (intact from the base knuckle to the shoulder)
* Intact skin on the dorsum of the hand, the ventral forearm, and antecubital fossa, without rash, irritation, scarring, open abrasion or other injury in these sites.
* Participant does not have an acute or critical medical illness or injury requiring immediate evaluation and/or treatment.

Exclusion Criteria

* Younger than 18 years of age
* No intact upper extremities
* The participant does not have intact skin on the dorsum of the hand, the ventral forearm, and antecubital fossa, without rash, irritation, scarring, open abrasion or other injury preventing appropriate evaluation of these sites.
* Non-English speaking participant.
* Patient has had current or recent (within 6 months) venous access in the arm that will be evaluated.
* Acute or critical illness or injury requiring immediate or urgent evaluation and treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric & Adult patients presenting at the Emergency Department that do not have an acute or critical medical illness or injury that required immediate evaluation and/or treatment.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-06; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of Veins Identified with VeinViewer will be greater than those identified by sight or sight & palpation | Immediately after assessment-Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Bruce M Becker, MD, Principal Investigator — Hasbro Children's Hospital
Locations (1):
- HASBRO Children's Hospital, Providence, Rhode Island, United States